CLINICAL TRIAL: NCT02721329
Title: Evaluation of APAP With SensAwake in OSA and Insomnia Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fisher and Paykel Healthcare (Industry)
Collaborators: University Hospital, Grenoble (Other); University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CIA-151; 2015-000407-57 (EudraCT Number)
Record Dates: First submitted 2016-03-23; First posted 2016-03-29 (Estimated); Last update posted 2020-07-02 (Actual); Status verified 2020-06

CONDITIONS: Obstructive Sleep Apnea; Insomnia
Keywords: Obstructive Sleep Apnea; OSA; Insomnia; CPAP; SensAwake
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- APAP without SensAwake (Active Comparator): Auto CPAP delivered from the ICON+ CPAP device.
  Interventions: Device: APAP
- APAP with SensAwake (Experimental): Auto CPAP with SensAwake turned on and set at a pressure of 4cmH2O. SensAwake is a pressure relief function that reduces the CPAP pressure on the transition from sleep to wake.
  Interventions: Device: APAP with SensAwake

INTERVENTIONS:
Device: APAP — Automatic Continuous Positive Airway Pressure
  Other Names: Automatic Continuous Positive Airway Pressure; Auto CPAP; ICON+ Auto
  Arms: APAP without SensAwake
Device: APAP with SensAwake — Automatic Continuous Positive Airway Pressure with SensAwake enabled. SensAwake is a pressure relief technology that detects the transition from sleep to wake, and promptly reduces the pressure during wakeful periods.
  Other Names: Automatic Continuous Positive Airway Pressure with SensAwake Pressure relief; ICON+ Auto with SensAwake Pressure relief; Auto CPAP with SensAwake Pressure relief
  Arms: APAP with SensAwake

SUMMARY:
The hypothesis is that APAP with SensAwake improves wake-after sleep onset compared to APAP without SensAwake in a patient population with Obstructive Sleep Apnea Syndrome (OSAS) and Insomnia.

DETAILED DESCRIPTION:
Patients with OSA and Insomnia will be enrolled into this randomized study to receive treatment with APAP with and without SensAwake. Baseline data will be collected for one week prior to CPAP initiation, followed by two treatment periods on each study arm of four weeks each.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years of age.
* Diagnosed with OSA and eligible for CPAP treatment under local requirements (AHI>30 with no more than 20% of central respiratory events)
* Naïve to CPAP therapy, i.e. have not been prescribed, or used CPAP in the last 5 years.
* Fluent in spoken and written French

Exclusion Criteria:

* Significant uncontrolled cardiac disease, as per the principal investigator's discretion, and/or Left Ventricular Ejection Fraction (LVEF) < 45%
* Co-existing lung disease, as per the principal investigator's discretion
* Co-existing sleep disorder, such as predominant central sleep apnea
* Previous or current diagnosis of sleep phase delay
* Pregnancy
* Participants that are unable or unwilling to give informed consent
* Receiving cognitive behavioral therapy or other intervention to treat insomnia. Subjects may be using hypnotics, but there shall be no change in hypnotic use during the protocol or 4 weeks preceding enrolment into the study.
* Diagnosed with clinical depression and/or currently using anti-depressants and/or anti-anxiolytics within the last 6 months.
* Hospital Anxiety OR Depression score > 11
* Participating in another research study for the duration of participation in this study. Participation in an observational study or genetic study is permitted at the discretion of the investigator.
* Patient protected by the Law, under guardianship or curators, as defined in Public Health Code in articles from L1121-5 to L1121-8.
* Patient not covered by a health insurance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2016-06; Primary Completion 2020-03 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
Objective Sleep Quality - Wake After Sleep Onset (WASO) | Four weeks
  Amount of time spent awake after sleep onset, as measured by actigraphy

SECONDARY OUTCOMES:
Objective Sleep Quality - Total Sleep Time | Four weeks
  Total sleep time, as measured by actigraphy - nightly average
Objective Sleep Quality - Sleep Onset Latency | Four weeks
  Time it takes to fall asleep, as measured by actigraphy - nightly average
Objective Sleep Quality - Sleep efficiency | Four weeks
  Percentage of time in bed spent asleep, as measured by actigraphy - nightly average
Treatment compliance | Four weeks
  Time spent on CPAP treatment - nightly average
Subjective sleep quality - Pittsburgh Sleep Quality Index | Four weeks
  Questionnaire
Insomnia severity - Insomnia Severity Index | Four weeks
  Questionnaire
Daytime sleepiness - Epworth Sleepiness Score | Four weeks
  Questionnaire
Quality of Life - Short Form 12 | Four weeks
  Questionnaire
Blood pressure | 24 hours
  Measured by 24 hour ambulatory blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Louis Pepin, MD, Principal Investigator — CHU du Grenoble
Locations (1):
- CHU Grenoble, Grenoble, France

IPD SHARING:
Plan to Share IPD: No